CLINICAL TRIAL: NCT00643344
Title: Craving and Lifestyle Management Through Mindfulness Pilot Study
Acronym: CALMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Mount Zion Health Fund (Other); Robert Deidrick Fund (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H7429-31882-01; Protocol 5030
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Obesity
Keywords: obesity; mindfulness based stress reduction; diet and exercise; mindful eating; stress
MeSH Terms: conditions — Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CALMM+ (Experimental): Participants receiving CALMM intervention, ie program that combines stress reduction, mindful eating practices with diet and exercise
  Interventions: Behavioral: Craving and Lifestyle Management through Mindfulness(CALMM+)
- TLC (Active Comparator): Participants receiving diet and exercise classes only
  Interventions: Behavioral: Craving and Lifestyle Management through Mindfulness(CALMM+)

INTERVENTIONS:
Behavioral: Craving and Lifestyle Management through Mindfulness(CALMM+) — MBSR is a program that provides systematic training in mindfulness meditation and gentle yoga as a self-regulation approach to reduce stress and improve medical and psychological symptoms. In this randomized controlled pilot study, we aim to test a 16-week intervention that further integrates diet and exercise into the CALMM program (CALMM+). This novel program, which includes elements drawn from MBSR, will be actively compared with the conventional diet and exercise group(TLC). Both groups will receive about 7 hours of in-class and out-of-class activities per week. The activities includes exercise, keeping dietary records, and stress reduction practices (if they are assigned to the intervention group).
  Other Names: CALMM2

SUMMARY:
The purpose of this study is to determine whether an innovative program that combines mindfulness-based stress reduction and mindful eating practices with diet and exercise guidelines (CALMM+ intervention) will lead to greater weight loss and more favorable body fat distribution than a conventional weight-loss program(Diet-Ex intervention).

DETAILED DESCRIPTION:
Obesity is an important growing epidemic, with about 65% of Americans overweight (Flegal, Carroll et al. 2002). Psychological stress is widely cited anecdotally as a factor that causes people to engage in overeating, and studies provide strong evidence that stress can promote obesity. Stress induces selective preference of sweet, high-fat food and increases visceral fat depots. Chronic stress has also been shown to impair immune responses, including decreasing immune responses to vaccination. The proposed study will pilot test an innovative program that combines stress reduction and mindful eating practices with diet and exercise, Craving and Lifestyle Management through Mindfulness (CALMM+). This program will be compared with diet and exercise intervention alone (Diet-Ex). Approximately 20 persons will be randomized to the two groups, which will meet weekly for 16 weeks. Key outcome measures are weight, fat distribution (as measured by waist/hip ratio), perceived stress, and mood. These measures will be assessed in visits performed at baseline, 3 months, and 6 months. Data from this study are intended to provide pilot data for use in planning a larger randomized, controlled trial that will compare the effects of the CALMM+ and Diet-Ex interventions on the metabolic and psychological processes assessed in this pilot study.

ELIGIBILITY:
Inclusion Criteria:

* healthy female
* aged 18-50
* BMI range 25-45
* negative urine glucose test
* must be able to provide informed consent

Exclusion Criteria:

* male
* age less than 18 or menopausal
* clinical diagnosis of eating disorder, diabetes, polycystic ovary syndrome, and coronary artery disease
* history of anginal chest pain without adequate evaluation
* substance abuse, mental health or medical condition that might interfere with study participation
* use of medications containing corticosteroids
* breastfeeding
* non- English speaker
* pregnant or planning to get pregnant in the next 6 months
* previous Mindfulness Based Stress Reduction training
* initiation of new class of psychiatric medications in past 2 months
* currently on a weight loss diet

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2008-01; Primary Completion 2008-10 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
weight | baseline, 3 month, and 6 month assessments

SECONDARY OUTCOMES:
fat distribution | baseline, 3 month, and 6 month assessments
perceived stress | baseline, 3 month, and 6 month assessments
mood | baseline, 3 month, and 6 month assessments

CONTACTS AND LOCATIONS:
Overall Officials: Frederick Hecht, MD, Principal Investigator — UCSF Osher Center for Integrative Medicine; Elissa Epel, PhD, Principal Investigator — UCSF Department of Psychiatry; Jennifer Daubenmier, PhD, Principal Investigator — UCSF Osher Center for Integrative Medicine
Locations (1):
- UCSF CTSI Clinical Research Center, San Francisco, California, United States

REFERENCES:
- [Background] Baer RA, Smith GT, Allen KB. Assessment of mindfulness by self-report: the Kentucky inventory of mindfulness skills. Assessment. 2004 Sep;11(3):191-206. doi: 10.1177/1073191104268029. PMID 15358875
- [Background] Flegal KM, Carroll MD, Ogden CL, Johnson CL. Prevalence and trends in obesity among US adults, 1999-2000. JAMA. 2002 Oct 9;288(14):1723-7. doi: 10.1001/jama.288.14.1723. PMID 12365955
- [Background] Epel ES, McEwen B, Seeman T, Matthews K, Castellazzo G, Brownell KD, Bell J, Ickovics JR. Stress and body shape: stress-induced cortisol secretion is consistently greater among women with central fat. Psychosom Med. 2000 Sep-Oct;62(5):623-32. doi: 10.1097/00006842-200009000-00005. PMID 11020091
- [Background] Dallman MF, Pecoraro N, Akana SF, La Fleur SE, Gomez F, Houshyar H, Bell ME, Bhatnagar S, Laugero KD, Manalo S. Chronic stress and obesity: a new view of "comfort food". Proc Natl Acad Sci U S A. 2003 Sep 30;100(20):11696-701. doi: 10.1073/pnas.1934666100. Epub 2003 Sep 15. PMID 12975524
- [Background] Oliver G, Wardle J, Gibson EL. Stress and food choice: a laboratory study. Psychosom Med. 2000 Nov-Dec;62(6):853-65. doi: 10.1097/00006842-200011000-00016. PMID 11139006
- [Background] Boggiano MM, Chandler PC, Viana JB, Oswald KD, Maldonado CR, Wauford PK. Combined dieting and stress evoke exaggerated responses to opioids in binge-eating rats. Behav Neurosci. 2005 Oct;119(5):1207-14. doi: 10.1037/0735-7044.119.5.1207. PMID 16300427
- [Background] Yusuf S, Hawken S, Ounpuu S, Bautista L, Franzosi MG, Commerford P, Lang CC, Rumboldt Z, Onen CL, Lisheng L, Tanomsup S, Wangai P Jr, Razak F, Sharma AM, Anand SS; INTERHEART Study Investigators. Obesity and the risk of myocardial infarction in 27,000 participants from 52 countries: a case-control study. Lancet. 2005 Nov 5;366(9497):1640-9. doi: 10.1016/S0140-6736(05)67663-5. PMID 16271645
- [Background] Epel E, Lapidus R, McEwen B, Brownell K. Stress may add bite to appetite in women: a laboratory study of stress-induced cortisol and eating behavior. Psychoneuroendocrinology. 2001 Jan;26(1):37-49. doi: 10.1016/s0306-4530(00)00035-4. PMID 11070333
- [Background] Epel E, Jimenez S, Brownell K, Stroud L, Stoney C, Niaura R. Are stress eaters at risk for the metabolic syndrome? Ann N Y Acad Sci. 2004 Dec;1032:208-10. doi: 10.1196/annals.1314.022. PMID 15677412
- [Background] Rebuffe-Scrive M, Walsh UA, McEwen B, Rodin J. Effect of chronic stress and exogenous glucocorticoids on regional fat distribution and metabolism. Physiol Behav. 1992 Sep;52(3):583-90. doi: 10.1016/0031-9384(92)90351-2. PMID 1409924
- [Background] Rosmond R. Role of stress in the pathogenesis of the metabolic syndrome. Psychoneuroendocrinology. 2005 Jan;30(1):1-10. doi: 10.1016/j.psyneuen.2004.05.007. PMID 15358437
- [Background] Roemmich JN, Wright SM, Epstein LH. Dietary restraint and stress-induced snacking in youth. Obes Res. 2002 Nov;10(11):1120-6. doi: 10.1038/oby.2002.152. PMID 12429875